CLINICAL TRIAL: NCT04708249
Title: D-chiroinositol Administration for Testosterone Level Improvement in Hypogonadal Males
Brief Title: D-chiroinositol Administration in Hypogonadal Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCI_HYPOGONADAL_MALES
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-01

CONDITIONS: Male Hypogonadism; Sexual Dysfunction
Keywords: Male Hypogonadism; Testosterone; Aromatase; D-chiroinositol; Sexual dysfunction
MeSH Terms: conditions — Eunuchism; Sexual Dysfunction, Physiological | interventions — kasugamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-chiroinositol treatment (Experimental)
  Interventions: Dietary Supplement: D-chiroinositol

INTERVENTIONS:
Dietary Supplement: D-chiroinositol — Supplementation with 600 mg of D-chiroinositol, two-times daily on an empty stomach, for 30 days.

SUMMARY:
D-chiroinositol (DCI), is known as second messenger of insulin pathway, but recently several works have reported the influence of DCI on steroidogenesis. In particular, the DCI capabilities to regulate aromatase expression and testosterone biosynthesis are arising. In this regard, DCI administration in case of reduced levels of testosterone, could be a good therapeutic opportunity. For this reason, the treatment of Late-Onset Male Hypogonadism (LOH) in undoubtedly an interesting target. LOH is a reduction of testosterone level due to advancing age, currently treated with Testosterone Replacement Therapy (TRT). Unfortunately, there is a lack of information about TRT safety, especially in older men. For these reasons, the aim of this study is to evaluate the effect of DCI treatment on testosterone accumulation in LOH patient.

ELIGIBILITY:
Inclusion Criteria:

* Men, with a diagnosis of Late-Onset Male Hypogonadism
* Insulin resistance (HOMA Index > 2,5)
* BMI between 25 and 30

Exclusion Criteria:

* Alcohol intake and/or drug abuse
* Recent hormonal treatment
* Smoking
* Obesity
* Systemic or endocrine diseases
* Male accessory gland infection
* Clinical history of cryptorchidism or varicocele and micro-orchidism

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Serum Testosterone at 1 month | At baseline and after 30 days of treatment
  Level of testosterone detected in the blood in ng/dL

SECONDARY OUTCOMES:
Change from Baseline Weight at 1 month | At baseline and after 30 days of treatment
  Body weight of patients reported in kg
Change from Baseline Waist circumference at 1 month | At baseline and after 30 days of treatment
  Waist circumference of patients reported in cm
Change from Baseline BMI at 1 month | At baseline and after 30 days of treatment
  Body Mass Index of patients calculated as kg/m2, where kg is the weight measured for eah patient while m2 is his height squared
Change from Baseline Insulin at 1 month | At baseline and after 30 days of treatment
  Level of fasting insulin detected in the blood and reported in microU/L
Change from Baseline Glycaemia at 1 month | At baseline and after 30 days of treatment
  Level of fasting glycaemia detected in the blood and reported in mg/dL
Change from Baseline HOMA index at 1 month | At baseline and after 30 days of treatment
  HOMA index known as Homeostatic Model Assessment for Insulin Resistance is: (fasting glycaemia x fasting insulin)/405
Change from Baseline Androstenedione at 1 month | At baseline and after 30 days of treatment
  Level of androstenedione detected in the blood and reported in ng/mL
Change from Baseline Luteinizing Hormone at 1 month | At baseline and after 30 days of treatment
  Level of luteinizing hormone detected in the blood and reported in mUI/ml
Change from Baseline Oestradiol at 1 month | At baseline and after 30 days of treatment
  Level of oestradiol detected in the blood and reported in pg/mL
Change from Baseline Oestrone at 1 month | At baseline and after 30 days of treatment
  Level of oestrone detected in the blood and reported in pg/mL
Change from Baseline Testosterone/Oestradiol ratio at 1 month | At baseline and after 30 days of treatment
  Ratio between the levels of oestradiol and testosterone detected in the blood
Change from Baseline Strength Test at 1 month | At baseline and after 30 days of treatment
  Measurement of strength performed with the dominant hand using a hand-held dynamometer (Good Strength, IGS01, Metitur Oy, Jyväskylä, Finland) with the participant in the seated position with elbow flexed at 110°. The participant will be instructed to squeeze the handle as hard as possible for 3-5 seconds and the stregth will be recorded in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alma Res, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nordio M, Kumanov P, Chiefari A, Puliani G. D-Chiro-Inositol improves testosterone levels in older hypogonadal men with low-normal testosterone: a pilot study. Basic Clin Androl. 2021 Nov 12;31(1):28. doi: 10.1186/s12610-021-00146-4. PMID 34763665